CLINICAL TRIAL: NCT03848650
Title: The Drift-Reduction for Improved Fractional Flow Reserve (FFR) Using Fiberoptic Technology (DRIFT) Study
Brief Title: The Drift-Reduction for Improved FFR Using Fiberoptic Technology (DRIFT) Study
Acronym: OPSENS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: AAAR7661
Record Dates: First submitted 2019-02-19; First posted 2019-02-21 (Actual); Results first posted 2024-06-11 (Actual); Last update posted 2024-06-11 (Actual); Status verified 2024-06

CONDITIONS: Left Anterior Descending Coronary Artery Stenosis
Keywords: FFR OCT LAD
MeSH Terms: interventions — Fractional Flow Reserve, Myocardial

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Opsens Medical OptoWire (Experimental): Subjects who will have or recently had FFR using the Opsens Medical OptoWire Deux FFR system.
  Interventions: Device: OpSens Medical OptoWire; Procedure: FFR

INTERVENTIONS:
Device: OpSens Medical OptoWire — The OptoWire is FDA approved to measure pressure in coronary vessels during diagnostic angiography and coronary interventions.
  The OptoWire Deux pressure wire (OpSens Medical, Quebec, Canada) is a novel technology utilizing optical coherence technology to enhance FFR assessment of the coronaries.
  Other Names: OpSens Medical OptoWire Deux FFR System
Procedure: FFR — A guide wire-based procedure that can accurately measure blood pressure and flow through a specific part of the coronary artery. FFR is done through a standard diagnostic catheter at the time of a coronary angiogram (a.k.a. cardiac catheterization).
  Other Names: Fractional Flow Reserve

SUMMARY:
The primary objective of this study is to assess the accuracy, efficacy, and durability of the OpSens Medical OptoWire Deux pressure wire in the assessment of angiographically intermediate proximal left anterior descending coronary artery (LAD) stenoses in clinical practice.

DETAILED DESCRIPTION:
This study is designed as a prospective, observational in nature, multi-center, single-arm, clinical registry to estimate the ischemic burden of angiographically intermediate proximal LAD stenosis in clinical practice using the OpSens Medical OptoWire Deux FFR system. Subjects with stable angina or unstable angina who are found to have an intermediate proximal LAD stenosis on coronary angiography with anatomy amenable to PCI and underwent physiological lesion assessment with the OptoWire Deux pressure wire and OCT as part of their routine procedures using standard of care techniques will be enrolled. Patients meeting enrollment criteria will be offered the opportunity to enroll in this observational registry post-procedure. All patients enrolled in this study are expected to be evaluated and treated using a standard of care technique. This study will enroll a total of 60 patients at Columbia University Medical Center and St. Francis Hospital.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects, >18 years of age.
* Patients with stable angina, unstable angina or non-ST segment elevation myocardial infarction (if the LAD lesion is the non-culprit lesion) and in whom an intermediate proximal LAD de novo stenosis (30-80%) with TIMI flow 3 has been identified on angiography. Note: Patients with multi-vessel disease can be enrolled.
* Patients have had fractional flow reserve (FFR) and optical coherence tomography (OCT) of the LAD with the OpSens FFR system as part of their routine evaluation as standard of care procedure.
* Provides written, informed consent and HIPAA consent to use the data in a clinical study.

Exclusion Criteria:

(General exclusion criteria)

* Patients presented with NSTEMI with the LAD involved as the culprit lesion
* Any ST-elevation myocardial infarction within the past 30 days.
* Hemodynamic instability requiring vasopressor or mechanical circulatory support.
* Prior heart transplant.
* Known left ventricular ejection fraction ≤40%.
* LAD supplying akinetic or severely hypokinetic territories if already known based on prior imaging.
* Patient is enrolled in another clinical study that may impact the results of this study.
* FFR not acquired per instructions for the OpSens Wire.
* LAD Lesion not assessed with OCT.

(Angiographic exclusion criteria)

* Thrombolysis in Myocardial Infarction (TIMI) grade 2 or lower at baseline angiography.
* Target lesion involves left main (stenosis >50%).
* Previous percutaneous coronary intervention (PCI) with stent in LAD or left main trunk.
* Presence of chronic total occlusion in any vessel.
* Presence of a side branch≥2.75 mm with ≥70% stenosis in the LAD.
* Bifurcation lesion that resulted in the stent implantation of a side branch.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2018-06-19 (Actual); Primary Completion 2019-05-13 (Actual); Study Completion 2019-05-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Manish Parikh, MD, Principal Investigator — Columbia University
Locations (2):
- United States (2):
  - New York Presbyterian Hospital/Columbia University Medical Center, New York, New York
  - St. Francis Hospital, Roslyn, New York

IPD SHARING:
Plan to Share IPD: No
We do not plan to share individual participant data (IPD) with other researchers.

RESULTS

PARTICIPANT FLOW:
Groups:
- Opsens Medical OptoWire: Subjects who will have or recently had Fractional Flow Reserve (FFR) using the Opsens Medical OptoWire Deux FFR system.
  OpSens Medical OptoWire: The OptoWire is FDA approved to measure pressure in coronary vessels during diagnostic angiography and coronary interventions.
  The OptoWire Deux pressure wire (OpSens Medical, Quebec, Canada) is a novel technology utilizing optical coherence technology to enhance FFR assessment of the coronaries.
  Fractional Flow Reserve (FFR): A guide wire-based procedure that can accurately measure blood pressure and flow through a specific part of the coronary artery. FFR is done through a standard diagnostic catheter at the time of a coronary angiogram (a.k.a. cardiac catheterization).
Period: Overall Study
Arm/Group | Opsens Medical OptoWire
Started | 60
Completed | 60
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Opsens Medical OptoWire: Subjects who will have or recently had FFR using the Opsens Medical OptoWire Deux FFR system.
  OpSens Medical OptoWire: The OptoWire is FDA approved to measure pressure in coronary vessels during diagnostic angiography and coronary interventions.
  The OptoWire Deux pressure wire (OpSens Medical, Quebec, Canada) is a novel technology utilizing optical coherence technology to enhance FFR assessment of the coronaries.
  FFR: A guide wire-based procedure that can accurately measure blood pressure and flow through a specific part of the coronary artery. FFR is done through a standard diagnostic catheter at the time of a coronary angiogram (a.k.a. cardiac catheterization).
Arm/Group | Opsens Medical OptoWire
Number analyzed (Participants) | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 65 (8.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18
  Male | 42
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 60
Hypertension [Count of Participants; unit: Participants] | 45

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Recordings of Significant Drift in Pre and Post-PCI
Description: The rate of significant drift is defined as FFR <0.97 or >1.03 with the in the pre-percutaneous coronary intervention (PCI) FFR recording using the OpSens OptoWire Deux pressure wire system. FFR is calculated by measuring the ratio between pressure distal to a stenosis and pressure proximally to stenosis using specialized pressure-measuring guidewires during maximal hyperemia.
Time Frame: During procedure, approximately less than an hour
Measure: Number; unit: Percentage
Units Other Than Participants: FFR recordings
Arm/Group | Opsens Medical OptoWire
Number analyzed (Participants) | 60
Number analyzed (FFR recordings) | 60
Percentage | 5.8

ADVERSE EVENTS:
Time Frame: During procedure, approximately up to 1 hour
Arm/Group | Opsens Medical OptoWire
All-Cause Mortality (participants affected / at risk) | 0/60
Serious Adverse Events (participants affected / at risk) | 0/60
Other Adverse Events (participants affected / at risk) | 0/60

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-11-20): https://cdn.clinicaltrials.gov/large-docs/50/NCT03848650/Prot_SAP_000.pdf